CLINICAL TRIAL: NCT04753177
Title: The Neoadjuvant Combined Hormone Therapy in Premenopausal Women With Locally Advanced ER+/HER2- Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint Petersburg State Budgetary Healthcare Institution, City Clinical Oncology Dispensary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2021-02-06; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: The Neoadjuvant Therapy
Keywords: combined hormone therapy; CDK4/6-ingibitors; fulvestrant; gozerelin; triptorelin
MeSH Terms: interventions — Fulvestrant; Triptorelin Pamoate; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant combined hormone therapy (Experimental): Ribocyclib, fulvestrant, triptorelin
  Interventions: Drug: Ribocyclib, fulvestrant, triptorelin; Drug: Doxorubicin, cyclophosphamide, paclitaxel
- Chemotherapy (the control) (Active Comparator): doxorubicin, cyclophosphamide, paclitaxel
  Interventions: Drug: Ribocyclib, fulvestrant, triptorelin; Drug: Doxorubicin, cyclophosphamide, paclitaxel

INTERVENTIONS:
Drug: Ribocyclib, fulvestrant, triptorelin — Neoadjuvant treatment will last 24 weeks in both groups. A follow-up examination will be carried out every 8 weeks. In the group of combined hormone therapy, repeate cor-biopsy of the tumor is planned to assess the Ki-67
Drug: Doxorubicin, cyclophosphamide, paclitaxel — Neoadjuvant treatment will last 24 weeks in both groups. A follow-up examination will be carried out every 8 weeks. In the group of combined hormone therapy, repeate cor-biopsy of the tumor is planned to assess the Ki-67

SUMMARY:
Breast cancer take a leading position in the structure of morbidity and mortality from malignant tumors among women.

Today the interest of many scientists and pharmaceutical companies is focused on the study of metastatic breast cancer forms. While we obtain little experimental data and practical research about the treatment of locally advanced forms.

In this regard, the study of new neoadjuvant drug therapy regimen for estrogen-receptor positive breast cancer in premenopausal woman is very relevant.

The proposed research will be the absolutely innovative investigation worldwide.

The study will consist of two modes of treatment, combined hormone therapy with CDK4/6-ingibitors and chemotherapy (the control), each replicated four times in a randomized, complete block design.

This research aims to improve the results of treatment, namely to increase the percentage of successfully treated patients and reduce toxicity from treatment.

Primary study endpoints will include the frequency of objective response and complete pathomorphological response (according to the Miller-Payne classification).

Secondary endpoints will include a decrease of the Ki67 level in postoperative material compared to primary biopsy, the frequency of organ-preserving operation after neoadjuvant treatment and quality of life.

Study hypothesis: neoadjuvant combined hormone therapy with CDK4/6-ingibitors in premenopausal women with luminal breast cancer leads to at least the same results as neoadjuvant chemotherapy, but with less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* Women with a newly diagnosed breast cancer who have not previously received specific treatment, with a tumor stage: cT1-3N1-2M0.
* Immunohistochemical tumor markers: ER-positive (ER+ is defined ≥ 10% and/or and Allred of 2 or more); HER2 negative (HER2 negative is defined as having an IHC of 1+ without ISH OR IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells OR ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)
* Premenopausal women.
* Signed consent to participate in a clinical trial.
* The consent of the patient to carry out, if possible, organ-preserving surgery with previous radiation therapy.
* General state of ECOG (PS) 0 or 1.
* Adequate Bone Marrow Function including:

Absolute Neutrophil Count (ANC) ≥1500/μL or ≥1.5 x109/L; Platelets ≥100000/μL or ≥100 x 109/L; Hemoglobin ≥ 9 g/dL.

* Adequate Renal Function including: Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution.
* Adequate Liver Function, including all of the following parameters:

Total serum bilirubin ≤ 1.0 x ULN unless the subject has documented Gilbert syndrome (in which case up to 3 x ULN is acceptable) ; Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN.

* Female subjects of child bearing potential and their partners, who are sexually active, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for at least 90 days after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse. Use of oral hormonal contraceptive agents in this study is not permitted.
* Absence of mutations in the BRCA1 and BRCA2 genes (revealed by PCR blood analysis)
* Providing histological materials to determine the status of mutations in the PIK3CA gene

Exclusion Criteria:

* Primary multiple synchronous tumors (except for detected basal multiple cancer of the skin or cervix in situ, which can be radically treated without adjuvant treatment for breast cancer)
* HIV positive status
* Known hypersensitivity to study drugs or excipients.
* Pregnancy and lactation
* Any chronic disease in the acute stage

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-01-28 (Estimated); Study Completion 2024-01-28 (Estimated)

PRIMARY OUTCOMES:
frequency of objective response | 24 weeks
  according to the results of ultrasound of the mammary glands and / or mammography
complete pathomorphological response | 24 weeks
  according to the Miller-Payne classification

SECONDARY OUTCOMES:
change of the Ki67 level in postoperative material compared to primary biopsy | 24 weeks
  compared to primary biopsy
the frequency of organ-preserving operation after neoadjuvant treatment | 24 weeks
  in bouth groups
quality of life | 24 weeks
  The quality of life questionnaire EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State Budgetary Healthcare Institution, City Clinical Oncology Dispensary, St-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
yes